CLINICAL TRIAL: NCT06502288
Title: Evaluation of Necessity of Antibiotic Administration Following Tooth Extraction: A Randomized Control Trial
Brief Title: Evaluation of Antibiotic Administration Following Tooth Extraction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chittagong Medical College (Other)
Responsible Party: Principal Investigator, Salim Uddin, Lecturer, Children Dentistry, Chittagong Medical College
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 59.27.0000.013.19.PG.2024/324
Record Dates: First submitted 2024-07-07; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Tooth Extraction
Keywords: Antibiotic, tooth extraction, RCT
MeSH Terms: interventions — Amoxicillin

STUDY DESIGN:
Intervention Model Description: Intervention Group-A: Administration of a specific antibiotic regimen post-extraction.
  Control Group-B: Administration of no antibiotic.
  For group A, patients will be prescribed 625 mg of amoxicillin with combined clavulanic acid tablets three times a day after meals for 7 days following extraction. For group B, no post-operative antibiotics will be administered. Both groups will be given a non-steroidal anti-inflammatory drug, 400 mg ibuprofen, and an H2 receptor blocker, 20 mg omeprazole, twice daily before meals.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The surgeon, patients and the outcome assessor will be blind for the duration of the study.
  Participants: After teeth extraction, participants receive either the antibiotic or not without knowing which one they take.
  Surgeon: The clinicians who prescribe and administer the medication will not know whether they are giving the antibiotic or not. This can be achieved by having a third-party individual prescribe and distribute the medications according to the randomization schedule.
  Outcome Assessor: The individual assessing the outcomes (e.g., infection rates, healing times) will also be blinded to which treatment the participant received. This prevents bias in the evaluation of the treatment effects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group-A: Administration of a specific antibiotic regimen post-extraction. (Experimental): Patients will be prescribed 625 mg of amoxicillin with combined clavulanic acid tablets three times a day after meals for 7 days following extraction and also a non-steroidal anti-inflammatory drug, 400 mg ibuprofen, and an H2 receptor blocker, 20 mg omeprazole, twice daily before meals.
  Interventions: Drug: 625 mg of amoxicillin with combined clavulanic acid tablet
- Control Group-B: Administration of no antibiotic. (No Intervention): No post-operative antibiotics will be administered, patients will be prescribed a non-steroidal anti-inflammatory drug, 400 mg ibuprofen, and an H2 receptor blocker, 20 mg omeprazole, twice daily before meals.

INTERVENTIONS:
Drug: 625 mg of amoxicillin with combined clavulanic acid tablet — The intervention group must take 625 mg of amoxicillin with combined clavulanic acid tablets three times a day after meals for 7 days following extraction.
  Other Names: Tablet. Bioclavid 625 mg
  Arms: Intervention Group-A: Administration of a specific antibiotic regimen post-extraction.

SUMMARY:
The trial aims to evaluate the effects of prescribing antibiotics after tooth extraction. 152 dental patients aged 18 to 50 will be randomly assigned. The study will assess infection rates, healing times, pain, and adverse effects in patients who receive antibiotics versus those who do not. The trial will be conducted at the Oral and Maxillofacial Surgery Department, Dental Unit, Chittagong Medical College. Data analysis will involve the use of the χ²-test, t-tests, and logistic regression, with a significance level of 5%. Ethical considerations include obtaining informed consent from all participants, and safety will be monitored by an independent expert team.

DETAILED DESCRIPTION:
Antibiotics are commonly prescribed in dentistry as a prophylactic measure, particularly following tooth extraction which are overused and misused in dental practice, leading to a rise in antimicrobial resistance. By randomly assigning 152 dental patients aged between 18 to 50 years, this trial aims to evaluate the outcomes such as infection rates, healing times, pain and adverse effects of patients receiving antibiotics after tooth extraction versus those who do not. The study will be conducted at the Oral and Maxillofacial Surgery Department, Dental Unit, Chittagong Medical College.

Tooth extractions will be performed under aseptic conditions, followed by standard post-operative care. The intervention group will receive 625 mg amoxicillin with clavulanic acid three times daily for 7 days post-extraction, while the control group will not receive any antibiotic. Both groups will receive 400 mg ibuprofen and 20 mg omeprazole twice daily. Surgeons, patients and assessors will be blinded to group assignments, with a third party managing medication distribution. Clinical evaluations will occur on the 3rd, 7th, and 14th days post-extraction. The Landry wound healing index will be used to assess tissue healing and pain will be recorded using a visual analogue scale. Surgical Site Infection will be diagnosed based on specific clinical criteria. Any Adverse reactions will be monitored. Rescue Additional analgesia and antibiotics will be provided as needed.

Data analysis will be done using the χ²-test, t-tests and logistic regression, with a significance level of 5%. Ethical considerations include obtaining informed consent from all participants. An independent expert team will conduct safety monitoring to manage any adverse events. The results of this study could provide valuable insights for future clinical protocols in dental surgery and contribute to the broader public health goal of reducing unnecessary antibiotic use.

ELIGIBILITY:
Inclusion Criteria:

1. Patient indicated extraction of teeth
2. Provide informed written consent
3. Patients aged between 18 to 50 years

Exclusion Criteria:

1. The tooth with abscess, infected cyst and tumors that require extensive surgery including impacted teeth
2. Patients who have taken antibiotics before 5 days for any reason will be excluded
3. Patients who are medically compromised such as DM, Congenital cyanotic heart disease, chronic kidney disease (CKD), Patients with chemotherapy or radiotherapy, Chronic Liver Disease (CLD), etc.
4. Female patients who are pregnant or lactating
5. Those women during the menstruation period (disturbed fibrinolytic activity),
6. Participants who are known hypersensitive to the given drugs used in this study
7. Participants who have known resistance to intervention drugs

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 152 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of post-extraction infections | 3rd, 7th, and 14th post-extraction day
  Surgical site infection will be diagnosed if the patient presents at least one of the following: A: Purulent drainage from the surgical wound or abscess. B: Isolation of pathogenic microorganisms in liquid or tissue cultures from the surgical site. C: Spontaneous opening of the incision site in patients with at least one of the following signs or symptoms: 1) fever (>38°C), 2) pain from palpation or spontaneous, 3) localized swelling, facial erythema or local heat. D: Severe pain after a week, together with moderate or severe inflammation or redness in the mouth and/or moderate or severe intraoral redness with no other apparent cause, that improves with antibiotic treatment.

SECONDARY OUTCOMES:
Healing time | 3rd, 7th, and 14th post-extraction day
  The Landry wound healing index will be used to assess the tissue healing process at the surgical sites. The assessment will involve evaluating specific parameters such as tissue color, bleeding response to palpation, the presence of granulation tissue, the characteristics of the incision margins, and the presence of suppuration on the 3rd, 7th, and 14th days after the operation. The index classifies the healing pattern based on the color of the soft tissue (pink or red), the presence or absence of suppuration, the amount of bleeding, the presence of granulation tissue, and the exposure of connective tissue into five different categories: (1) very poor, (2) poor, (3) good, (4) very good, and (5) excellent
Pain perception | 3rd, 7th, and 14th post-extraction day
  Pain perception of the patients will be measured using a visual analogue scale (VAS) ranging from 0 (no pain) to 10 (excessive pain) on the follow-up days
Adverse reaction | 3rd, 7th, and 14th post-extraction day
  We also evaluate adverse reactions related to the use of antibiotics, defined as follows: 1) Allergic reaction: urticaria and/or angioedema, 2) Anaphylaxis: throat or tongue swelling and/or respiratory symptoms. 3) Gastrointestinal reactions: nausea, vomiting, abdominal pain and diarrhea

CONTACTS AND LOCATIONS:
Overall Officials: Md Salim Uddin, BDS, MPhil, Principal Investigator — Chittagong Medical College
Locations (1):
- Chittagong Medical College, Chittagong, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
The study protocol will be available
Supporting Information: Study Protocol
Time Frame: August 15, 2025 to August 30, 2025
Access Criteria: Researchers interested
URL: http://clinicaltrials.gov/